CLINICAL TRIAL: NCT03691402
Title: A Randomized Controlled Trial Examining the Efficacy of Metacognitive Training for Depression in Later Life (MCT-Silver)
Brief Title: Evaluation of Metacognitive Training for Depression in Later Life (MCT-Silver)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Prof Dr. Steffen Moritz, Professor; Head of AG Clinical Neuropsychology, Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LPEK-005
Record Dates: First submitted 2018-09-25; First posted 2018-10-01 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Cognitive Remediation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MCT-Silver (Experimental): Metacognitive training for depression in later life is a cognitive-behaviorally based group therapy, which focuses on helping participants gain (metacognitive) distance from their thought patterns that contribute to depression. Over 8 modules, MCT-Silver addresses issues specific to depression in later life, such as coping with physical changes and loss, as well as adapting to new (social) roles. The program also includes modules on identifying and (re-)defining values in later life and how one may move toward acceptance of situations that cannot be prevented or changed. MCT-Silver addresses cognitive and metacognitive biases that contribute to the onset and maintenance of depression through fun and engaging exercises, as well as using examples from daily life.
  Interventions: Behavioral: MCT-Silver
- Cognitive Remediation (Active Comparator): mybraintraining© is a computer-based cognitive remediation program, which covers a wide range of neuropsychological exercises involving memory, reasoning, selective attention and psychomotor speed. The program is administered individually on personal computers and each session lasts approximately 45-60 min. To match the MCT-Silver group, participants will complete up to eight sessions of cognitive remediation.
  Interventions: Behavioral: Cognitive Remediation

INTERVENTIONS:
Behavioral: MCT-Silver — Metacognitive training for depression in later life (MCT-Silver) is a cognitive-behaviorally based group therapy, which focuses on helping participants gain (metacognitive) distance from their thought patterns that contribute to depression. Over 8 modules, MCT-Silver addresses issues specific to depression in later life, such as coping with physical changes and loss, as well as adapting to new (social) roles. The program also includes modules on identifying and re-defining values in later life and how one may move toward acceptance of situations that cannot be prevented or changed. MCT-Silver addresses cognitive and metacognitive biases that contribute to the onset and maintenance of depression through fun and engaging exercises, as well as using examples from daily life.
  Arms: MCT-Silver
Behavioral: Cognitive Remediation — mybraintraining© is a computer-based cognitive remediation program, which covers a wide range of neuropsychological exercises involving memory, reasoning, selective attention and psychomotor speed. The program is administered individually on personal computers and each session lasts approximately 45-60 min. To match the MCT-Silver group, participants will complete up to eight sessions of cognitive remediation.
  Arms: Cognitive Remediation

SUMMARY:
The study will evaluate the efficacy of metacognitive training for depression in later life (MCT-Silver) vs. cognitive remediation (mybraintraining©) in reducing depressive symptoms among older adults.

DETAILED DESCRIPTION:
The study examines the efficacy of Metacognitive Training for depression in later life (MCT-Silver). The study intends to investigate the extent to which MCT-Silver leads to a significant reduction in depressive symptoms compared to an active control group (mybraintraining©) (primary outcome: change in clinician-assessed depressive symptoms from t0 to t1 and t2). Secondary outcomes include change in self-reported depressive symptoms and dysfunctional (meta) cognitive beliefs, as well as quality of life, rumination, self-reported anxiety, attitudes toward aging and neuropsychological functioning from t0 to t1 and t2. The study design is a randomized-controlled trial with one intervention group and one active control group.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent
* age 60 years or older
* diagnosis of a single episode or recurrent major depressive disorder (MDD) or dysthymia (verified by the MINI)
* sufficient command of the German language
* willingness to participate in intervention over a period of 8 weeks (participants who do not attend the intervention will also be included in the analysis)
* Visual and auditory acuity adequate for neuropsychological testing and participation in group sessions

Exclusion Criteria:

* lifetime psychotic symptoms (i.e., hallucinations, delusions or mania)
* acute suicidal tendency
* intellectual disability (estimated IQ < 70)
* dementia or other neurological illness

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-11-18 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HRSD-24) | Total Time Frame is 5 months. Outcome is assessed at two points: baseline to post-assessment (8 weeks) and baseline to follow-up (5 months)
  The 24-item version of the Hamilton Depression Rating Scale is an established clinician-rated assessment of depressive symptom severity and assesses psychological as well as somatic symptoms (scores range from 0-2 or 0-4) of depression. The clinician rates the severity of these symptoms based on the patient's report and his or her own observation. Scores range from 0-54. Based on the first 17 items, a score of 8-13 indicates mild depression, 14-18 indicates moderate depression, 19-22 indicates severe depression and scores greater than 23 indicate very severe depression. The scale has demonstrated good sensitivity and specificity among older adults (Mottram, Wilson & Copeland, 2001). The reliability and validity among older adult samples has also been confirmed (Korner et al., 2006). In terms of assessing change for the current trial, a greater reduction in depressive symptoms (i.e., change score) indicates better outcome.

SECONDARY OUTCOMES:
16-item Quick Inventory for Depression (QIDS-C16) | Total Time Frame is 5 months. Outcome is assessed at two points: baseline to post-assessment (8 weeks) and baseline to follow-up (5 months)
  Change in rater-assessed depression as measured by the 16-item Quick Inventory for Depression (QIDS-C16) total score from baseline to post-assessment (8 weeks) and baseline to follow-up (5 months). Total scores range from 0-27 with higher scores indicating more severe levels of depression.
Beck Depression Inventory (BDI) | Total Time Frame is 5 months. Outcome is assessed at two points: baseline to post-assessment (8 weeks) and baseline to follow-up (5 months)
  Change in self-assessed depression as measured by the Beck Depression Inventory (BDI) total score from baseline to post-assessment (8 weeks) and baseline to follow-up (5 months). The BDI is a 21-item self-report measure of depression symptoms. Total scores range from 0-63 with higher scores indicating more severe levels of depression.
Dysfunctional Attitudes Scale Form 18B (DAS-18B) | Total Time Frame is 5 months. Outcome is assessed at two points: baseline to post-assessment (8 weeks) and baseline to follow-up (5 months)
  Change in dysfunctional attitudes as measured by change in the Dysfunctional Attitudes Scale Form 18B (DAS-18B) total score and subscale scores from baseline to post-assessment (8 weeks) and baseline to follow-up (5 months). Each item is endorsed on a 7-point scale (Range: 0-7) such that a total score of 126 is possible with higher scores indicating dysfunctional beliefs which are held more strongly. The total score is comprised of two subscales (perfectionism (Range 0-56); need for social approval (Range 0-21)), which are summed along with 7 other items to calculate the total scale score.
Metacognitions Questionnaire (MCQ-30) | Total Time Frame is 5 months. Outcome is assessed at two points: baseline to post-assessment (8 weeks) and baseline to follow-up (5 months)
  Change in metacognitive beliefs as measured by change in the Metacognitions Questionnaire (MCQ-30) total score and subscale scores from baseline to post-assessment (8 weeks) and baseline to follow-up (5 months). The 30-item scale has a range of 30-120. The scale is comprised of five subscales (range for each = 6-24): (1) Positive Beliefs (PB) about worry (6 items); (2) Negative Beliefs (NB) about thoughts concerning uncontrollability and danger (6 items), and (3) beliefs about the need to control thoughts (Need for Control [NFC],6 items); (4) Cognitive Confidence (6 items) and Cognitive Self-Consciousness (6 items). Higher scores indicate more strongly held metacognitive beliefs.
Rosenberg Self-Esteem Scale | Total Time Frame is 5 months. Outcome is assessed at two points: baseline to post-assessment (8 weeks) and baseline to follow-up (5 months)
  Change in self-esteem as measured by change in the Rosenberg Self-Esteem scale total score from baseline to post-assessment (8 weeks) and baseline to follow-up (5 months). The scale is comprised of 10 items and scores range from 10-40 with higher scores indicating higher self-esteem.
Ruminative Responses Scale | Total Time Frame is 5 months. Outcome is assessed at two points: baseline to post-assessment (8 weeks) and baseline to follow-up (5 months)
  Change in rumination as measured by the Ruminative Responses Scale total score from baseline to post-assessment (8 weeks) and baseline to follow-up (5 months). The scale is comprised of 10 items and scores range from 10-40 with higher scores indicating higher self-esteem.
World Health Organization Quality of Life-BREF - Item 1 | Total Time Frame is 5 months. Outcome is assessed at two points: baseline to post-assessment (8 weeks) and baseline to follow-up (5 months)
  Change in global quality of life as measured by change on item 1 on the World Health Organization Quality of Life-BREF from baseline to post-assessment (8 weeks) and baseline to follow-up (5 months). Responses on the item range from 1 (very bad quality of life) to 5 (very good quality of life).
Remission rate | Total Time Frame is 5 months. Outcome is assessed at two points: baseline to post-assessment (8 weeks) and baseline to follow-up (5 months)
  Remission rate at post-assesment (8 weeks) and follow-up (5 months) as measured by the Hamilton Depression Rating Scale (HDRS score ≤ 8)
EurQoL Group 5Q 5D 5L | Total Time Frame is 5 months. Outcome is assessed at two points: baseline to post-assessment (8 weeks) and baseline to follow-up (5 months)
  Change in health status as assessed by change in percentage of participants experiencing health-related difficulties in 5 domains and change in overall health quality as assessed by change on the Visual Analogue rating Scale (VAS; range 0-100; higher scores indicate better quality of life) from baseline to post-assessment (8 weeks) and baseline to follow-up (5 months).
Trail-Making Test, Part B | Total Time Frame is 5 months. Outcome is assessed at two points: baseline to post-assessment (8 weeks) and baseline to follow-up (5 months)
  Change in executive functioning as measured by change in the Trail-Making Test, Part B (TMT-B) time to completion from baseline to post-assessment (8 weeks) and baseline to follow-up (5 months). A maximum of 300 seconds is allowed and shorter time indicating better performance.
Trail-Making Test, Part A | Total Time Frame is 5 months. Outcome is assessed at two points: baseline to post-assessment (8 weeks) and baseline to follow-up (5 months)
  Change in Information processing speed as measured by change in the the Trail-Making Test A (TMT-A) time to completion from baseline to post-assessment (8 weeks) and baseline to follow-up (5 months). A maximum of 300 seconds is allowed and shorter time indicating better performance.
Rivermead Behavioral Memory Test | Total Time Frame is 5 months. Outcome is assessed at two points: baseline to post-assessment (8 weeks) and baseline to follow-up (5 months)
  Change in memory functioning as measured by change in Rivermead Behavioral Memory Test (RBMT) total score from baseline to post-assessment (8 weeks) and baseline to follow-up (5 months). Total scores range from 0-24 with higher scores indicating better memory performance.
Stroop Color-Word Task | Total Time Frame is 5 months. Outcome is assessed at two points: baseline to post-assessment (8 weeks) and baseline to follow-up (5 months)
  Change in executive functions as measured by the Stroop Color-Word test from baseline to post-assessment (8 weeks) and follow-up (5 months). The Stroop Color-Word test is comprised of three trials: Word Reading, Color Naming and Color-Word (CW) Naming. Per the Golden administration guidelines, total score for each subscale is the number of items completed within 45 seconds. For each condition, a raw score of 100 is possible (with a higher score indicating a better performance). For the current study, the Interference score will also be calculated, which is the difference between the expected CW Naming score and the predicted CW Naming score (which is predicted based on age and education; range is -29 to 30 such that larger scores indicate better performance).

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Moritz, PhD, Principal Investigator — Universtitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schneider BC, Veckenstedt R, Karamatskos E, Scheunemann J, Moritz S, Jelinek L, Miegel F. Change in negative mental filter is associated with depression reduction in metacognitive training for depression in older adults (MCT-Silver). Sci Rep. 2024 Jul 25;14(1):17120. doi: 10.1038/s41598-024-67063-0. PMID 39054326